CLINICAL TRIAL: NCT06709118
Title: The Effect of Different Fiberoptic Outer Diameters on Fiberoptic Intubation
Status: Not yet recruiting | Type: Observational
Sponsor: Qinye Shi (Other)
Responsible Party: Sponsor-Investigator, Qinye Shi, The Fourth Affiliated Hospital of Zhejiang University Medical College, The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Organization: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Other Study IDs: KY-2024-172
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Intubation Times
Keywords: Intubation; Ffiberoptic; Perioperative; Sore throat; Success rate
MeSH Terms: conditions — Pharyngitis | interventions — Optical Fibers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- 3.8mm Group: Orotracheal intubation was performed with a 3.8 millimeter outer diameter fiberoptic
  Interventions: Device: fiberoptic
- 2.8 mm group: Orotracheal intubation was performed with a 2.8 millimeter outer diameter fiberoptic
  Interventions: Device: fiberoptic
- 4.8mm group: Orotracheal intubation was performed with a 4.8 millimeter outer diameter fiberoptic
  Interventions: Device: fiberoptic

INTERVENTIONS:
Device: fiberoptic — Tracheal intubation was performed with different outer diameters of fiberoptic.

SUMMARY:
Fiberoptic intubation is an important method for anesthesiologists to deal with difficult airways, but its operation is difficult and requires repeated practice. Fiberoptic intubation is performed in two steps. First, the anesthesiologist holds the bronchoscope and exposes the base of the tongue, the epiglottis, and the glottis successively according to the front camera of the bronchoscope. Through the glottis, the main trachea is exposed to the carina. This process is visual and the anesthesiologist can see the main tissue structure directly. Then, the endotracheal catheter enters the endotracheal along the bronchoscope, and the process of endotracheal catheter entry is not visual.

In clinical work, it was found that the tracheal catheter was easily blocked when it passed through the glottis, and it was necessary to adjust the position of the tracheal catheter for several times before the tracheal catheter could be sent into the tracheal tube, which was easy to cause throat injury in the process. At present, relevant studies are mainly focused on the first step of bronchoscopic intubation, how to quickly expose the glottis and complete the bronchoscopic guidance process. However, there is no clear mention of the situation of catatoning in the process of endotracheal catheter and how to solve the problem of catatoning.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria，collecting the data of participants who undergone fiberoptic intubation. The observer analysis the safety and efficiency of fiberoptic intubation.

ELIGIBILITY:
Inclusion Criteria:

1.American Society of Anesthesiologists 1~2

2.18-60 year

3.Adult patients requiring general anesthesia for orotracheal intubation

Exclusion Criteria:

1. Limited mouth opening
2. limited movement of temporomandibular joint
3. abnormal glottic anatomy
4. polyps of vocal cords

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients in need of oral tube intubation and general anesthesia in our hospital for elective surgery
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Fiberoptic intubation attempts | during the procedure
  This is used to observe the passage of the tracheal tube through the glottis
First intubation success rate | during the procedure
  The incidence of tracheal tube through the vocal cords
Fiberoptic intubation time | during the procedure
  The duration of the intubation process
Time of passage of tracheal intubation through glottis | during the procedure
  The time the tracheal tube enters the trachea

SECONDARY OUTCOMES:
Hoarseness after surgery | 24 hours after surgery
  Patients were asked about voice changes 24 hours after surgery
Sore throat | 24 hours after surgery
  Patients were asked about throat pain 24 hours after surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piegeler T, Clausen NG, Weiss M. Effectiveness of tip rotation in fibreoptic bronchoscopy under different experimental conditions: an in vitro crossover study. Br J Anaesth. 2017 Dec 1;119(6):1206-1212. doi: 10.1093/bja/aex322. PMID 29028928
- [Background] Karmali S, Rose P. Tracheal tube size in adults undergoing elective surgery - a narrative review. Anaesthesia. 2020 Nov;75(11):1529-1539. doi: 10.1111/anae.15041. Epub 2020 May 16. PMID 32415788
- [Background] Teulieres M, Berard E, Marot V, Reina N, Ferre F, Minville V, Cavaignac E. A quadruple peripheral nerve block outside the OR for anterior cruciate ligament reconstruction reduces the OR occupancy time. Knee Surg Sports Traumatol Arthrosc. 2023 Jul;31(7):2917-2926. doi: 10.1007/s00167-022-07246-2. Epub 2022 Dec 5. PMID 36469051